CLINICAL TRIAL: NCT02952118
Title: Nasal Appliance for the Treatment of Snoring in Adult Subjects - A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GE Sleeping (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GES-ST-02-100
Record Dates: First submitted 2016-10-25; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one night with the device and one night without the device. (Experimental): The study duration with each patient will be 48 hours (two nights); at the first night the sleep study will be with PAT device, with snoring recording and without the "Forrest" epic device. In the second night the sleep study will be with PAT device, with snoring recording and with the "Forrest" epic device. The order of the sleep studies (with and without the epic device) will be randomly determined by computerized ahead prepared list. The research duration for patients that did not have a sleep study over the last year, will take place for 3 nights; the sleep study will be performed in order to make sure the patient does not suffer from obstructive respiratory disorder during sleep. The sleep studies will take place in a sleep laboratory (Millennium Sleep Labs LTD, Beer Sheva) or as an ambulatory study, at home.
  Interventions: Device: Forrest Snoring device

INTERVENTIONS:
Device: Forrest Snoring device

SUMMARY:
This is an open, pilot study for adults ( age range of 20-70 years old), who suffer from snoring without obstructive sleep apnea (OSA) and no need for CPAP treatment: with standard diagnosis of sleep study or with minor sleep disorder (AHI of less than 15 events per hour). Patients with no OSA over the last year will sign an informed consent after receiving explanations from authorized physician (Professor Asher Tal). The patient will than undergo a sleep study using a mobile device PAT (Peripheral Arterial Tomography, Itamar Medical, Israel) ,an approved device in Israel, USA and many other European countries,, approved for use by the USA FDA). This sleep study is needed in order to rule out OSA, namely AHI of more than 15 events per hour of sleep.

The study duration with each patient will be 48 hours (two nights); at the first night the sleep study will be with PAT device, with snoring recording and without the "Forrest" epic device. In the second night the sleep study will be with PAT device, with snoring recording and with the "Forrest" epic device. The order of the sleep studies (with and without the epic device) will be randomly determined by computerized ahead prepared list. The research duration for patients that did not have a sleep study over the last year, will take place for 3 nights; the sleep study will be performed in order to make sure the patient does not suffer from obstructive respiratory disorder during sleep. The sleep studies will take place in a sleep laboratory (Millennium Sleep Labs LTD, Beer Sheva) or as an ambulatory study, at home.

Recordings over the nights with or without the "Forrest" epic device will be carried out at the patient's home, after verification that each patient sleeps alone in his/her room. The recording and data processing of snoring will be performed through the application "SNORLAB" on IPHONE 6 mobile device. Ambulatory sleep studies with PAT device will be carried out during two nights (with and without the Forrest Device) with most patients.

During the examination, respiratory index will be tested such as: obstructive respiratory events during sleep, oxygen saturation in blood at rest (measured non-invasively) during sleep: mean, lowest (nadir), and rate of time the patient sleeps in with less than 90% of oxygen saturation in blood.

ELIGIBILITY:
Inclusion Criteria:

* The patient age range : 20-70 years old.
* The patient / legal guardian able and willing to sign conscious written agreement.
* The patient / legal guardian able and willing to comply with the study protocol.
* The patient is suffering from snoring.
* The patient underwent a sleep study over the last year.

Exclusion Criteria:

* The patient suffers from sleep apnea that requires CPAP treatment: more than 15 AHI per hour in a sleep study or due to significant background diseases.
* Patient less than 20 years old.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Difference between the two following parameters: (1) Total time of snoring during sleep with the device ("Forest") (2) Total time of snoring during sleep without the device. Resulting value is in minutes. | 1 year

SECONDARY OUTCOMES:
Snoring intensity at its peak, measured in decibels (dB). Resulting value is a number measured in dB Snoring intensity at its peak, measured in decibels (dB). Resulting value is a number measured in dB | 1 year
Number of obstructive events during sleep. Resulting value is an absolute number. | 1 year
Difference between the two following parameters: (1) Average oxygen saturation level with the device ("Forest") (2) Average oxygen saturation level without the device. Resulting value is in percents (%). | 1 year
Total time during which the oxygen saturation level is less than 90% during sleep with and without the device. Resulting value is in minutes | 1 year
Questionnaire: user experience (subjective) after a night with and without the device. Verbal description without scaling satisfaction. | 1 year